CLINICAL TRIAL: NCT07327255
Title: A Phase I, Randomized, Cross-over, Single-Center, Single Dose Fasted Study of EG-101 IV Injection (EG-ZNMP-01) in Healthy Volunteers to Serve as a Safety Lead-In for Dosing in Pregnant Women With Severe Pre-eclampsia
Brief Title: Pharmacokinetic Study to Evaluate Safety and Tolerability of EG-101 in Healthy Female Volunteers as a Safety Lead-In for Dosing in Pregnant Women With Severe Pre-eclampsia
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Evergreen Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: EG-101-1.1
Record Dates: First submitted 2025-12-02; First posted 2026-01-08 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-12

CONDITIONS: Pre-eclampsia
Keywords: Phase 1 Study
MeSH Terms: conditions — Pre-Eclampsia

STUDY DESIGN:
Intervention Model Description: Randomized, Cross-over, Single-Center, Single Dose Fasted Study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Group 1: treatment sequences ABC+D (Experimental): Period 1
  Drug: EG-101 100 mg IVPB once (Level A)
  Period 2
  Drug: EG-101 400 mg IVPB once (Level B)
  Period 3
  Drug: EG-101 600 mg IVPB once (Level C)
  Period 4
  Drug: EG-101 600 mg IVPB twice, 8 hours apart (Level D)
  Interventions: Drug: EG-101
- Group 2: treatment sequence: BCA+D (Experimental): Period 1
  Drug: EG-101 400 mg IVPB once (Level B)
  Period 2
  Drug: EG-101 600 mg IVPB once (Level C)
  Period 3
  Drug: EG-101 100 mg IVPB once (Level A)
  Period 4
  Drug: EG-101 600 mg IVPB twice, 8 hours apart (Level D)
  Interventions: Drug: EG-101
- Group 3: treatment sequence: CAB+D (Experimental): Period 1
  Drug: EG-101 600 mg IVPB once (Level C)
  Period 2
  Drug: EG-101 100 mg IVPB once (Level A)
  Period 3
  Drug: EG-101 400 mg IVPB once (Level B)
  Period 4
  Drug: EG-101 600 mg IVPB twice, 8 hours apart (Level D)
  Interventions: Drug: EG-101

INTERVENTIONS:
Drug: EG-101 — EG-ZNMP-01 IV injection 10 mg/mL, 20 mL vial
  Other Names: EG-ZNMP-01

SUMMARY:
Preeclampsia is one of the leading causes of maternal and fetal death. It is a syndrome of pregnant women and is usually characterized by new onset of hypertension and proteinuria after 20 weeks of gestation. This disease is a multisystem disorder affects most maternal organs, predominantly the vascular, renal, hepatic, cerebral and coagulation systems. While hypertension is almost always a symptom of this disease, preeclampsia is not the same as essential hypertension.

This is a single-center, randomized, open-label, 4 period, 3-way crossover, single dose fasted study to evaluate the safety, tolerability and pharmacokinetics of four ascending doses of the EG-101 IV injection in healthy volunteers.

Twenty-four subjects in total, with eight subjects randomly assigned to one of three different sequences for variation of doses under fasted conditions. Dosing duration is approximately 4 weeks and followed by the follow-up for each subject.

ELIGIBILITY:
Key Inclusion Criteria:

1. Healthy adult female volunteers, 18 to 55 years of age, inclusive, at first Check-In Visit
2. Body mass index (BMI) ≥18.5 to ≤32 kg/m2 at Screening (calculated as a function of measured height and weight according to the formula, BMI = kg / m2 where m2 is height in meters squared.)
3. All female subjects must be nonpregnant, nonlactating and either postmenopausal, surgically sterile, or using contraceptive regimens more than 3 months. All females must have a negative serum pregnancy test at Screening and Check-in Visit. Effective methods of contraception include a dual method of contraception: condom with spermicide in conjunction with use of an intrauterine device (IUD), condom with spermicide in conjunction with use of a diaphragm, condom with birth control patch or vaginal ring, or condom with oral, injectable, or implanted contraceptive. Surgical sterility is documented through documented: hysterectomy, partial hysterectomy, bilateral oophorectomy, or bilateral tubal ligation at least 6 months prior to Screening. Postmenopausal sterility is documented by absence of menses for at least 12 months prior to Screening plus serum FSH ≥40 mIU/mL and estradiol <30 pg/mL at screening
4. Male subjects, are not enrolled into this study
5. Medically healthy on the basis of medical history, and physical examination (including but not limited to an evaluation of the cardiovascular, gastrointestinal, respiratory, and central nervous systems), as determined by the Investigator at Screening and each Check-In Visit

Key Exclusion Criteria:

1. Females who are pregnant, lactating, or likely to become pregnant during the study
2. History and/or recent evidence within 6 months prior to Screening of alcohol or drug/substance abuse disorder
3. Subjects with a history of hypersensitivity to Zanamivir or any component of study medication
4. History of clinically significant allergies including drug allergies or allergic bronchial asthma or related bronchospastic conditions
5. Subjects who have history of unexplained syncope or fainting or a condition that predisposes them to syncope, such as hypotension, orthostatic hypotension, bradycardia or dehydration

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — The study enrolls only biological females and will accept only cisgender women.
Enrollment: 24 (Estimated)
Dates: Start 2026-06 (Estimated); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Tmax | Day 1 pre-dose and at multiple timepoints (up to 32 hours) post-dose
  Time to Maximum Concentration
Cmax | Day 1 pre-dose and at multiple timepoints (up to 32 hours) post-dose
  Maximum Plasma Concentration
AUC | Day 1 pre-dose and at multiple timepoints (up to 32 hours) post-dose
  Area Under the Plasma Concentration-time Curve
CL/F | Day 1 pre-dose and at multiple timepoints (up to 32 hours) post-dose
  Apparent Plasma Clearance
Vd/F | Day 1 pre-dose and at multiple timepoints (up to 32 hours) post-dose
  Apparent Volume of Distribution
t½ | Day 1 pre-dose and at multiple timepoints (up to 32 hours) post-dose
  Terminal Elimination Half-life
Ae | Day 1 pre-dose and at multiple timepoints (up to 32 hours) post-dose
  Cumulative Amount Excreted Unchanged in Urine

SECONDARY OUTCOMES:
Incidence of reported adverse events | From baseline through to post study Follow-up (up to 5 weeks)
  To assess the safety and tolerability of EG-101 across 4 ascending dose levels under fasting conditions in healthy women including but not limited to the adverse events.
Blood pressure | From screening throughout the study duration to post study Follow-up (up to 5 weeks)
Respiratory rate | From screening throughout the study duration to post study Follow-up (up to 5 weeks)
Pulse rate | From screening throughout the study duration to post study Follow-up (up to 5 weeks)
Body temperature | From screening throughout the study duration to post study Follow-up (up to 5 weeks)
12-lead electrocardiograms (ECG) | At the screening day, Day 1 pre-dose and 6 hours post-dose
  To assess the safety and tolerability of EG-101 across 4 ascending dose levels under fasting conditions in healthy women including but not limited to the resting 12-lead electrocardiograms (ECG) assessment (includes the overall interpretation, PR interval, QRS duration, RR, QT, and QTcF intervals).
Prothrombin time (PT) | On screening day, check-in day (D-1), and during post study Follow-up (up to 5 weeks)
  Clinical laboratory test of blood coagulation
White Blood Cell count | On screening day, check-in day (D-1), and during post study Follow-up (up to 5 weeks)
  Clinical laboratory test of hematology
Albumin | On screening day, check-in day (D-1), and during post study Follow-up (up to 5 weeks)
  Clinical laboratory test of serum chemistry
Protein | On screening day, check-in day (D-1), and during post study Follow-up (up to 5 weeks)
  Clinical laboratory test of urinalysis